CLINICAL TRIAL: NCT01289860
Title: A Controlled, Cross-over, Acute Intervention Study Investigating the Cognitive and Neuronal Effects of Flavonoids in Blueberries.
Brief Title: Investigating the Acute Effects of Flavonoids in Blueberries on Cognitive Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor of Nutritional Medicine, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UReading_2010_01
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Healthy Adults.
MeSH Terms: interventions — Flavonoids; Anthocyanins; Flavonols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blueberry drink (Active Comparator): 30g of blueberry powder (equivalent to 200g fresh blueberries) and 300ml of semi-skimmed milk
  Interventions: Dietary Supplement: Flavonoids
- Control drink (Placebo Comparator): 29g of powder consisting of sugars and vitamin C, values of which were matched to that of the blueberry drink, with 1 g of citric acid to match for taste.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Flavonoids — 475g of anthocyanidins in 300ml of blueberry drink.
  Other Names: Anthocyanidins, flavanols, flavonols.
  Arms: Blueberry drink
Dietary Supplement: Control — 29g powder: sugars (glucose, sucrose, fructose), vitamin C and citric acid.
  Arms: Control drink

SUMMARY:
This study was a controlled, cross-over, acute flavonoid intervention trial with younger and older adults. Subjects consumed a blueberry beverage during one visit and a control beverage on another. Cognitive function pre drink was assessed, blood and urine samples were taken as well as blood pressure and a measure of vascular reactivity. These outcome measures were taken at 2 and 5 hours post drink.

It was predicted that the flavonoids in the blueberry drink would lead to improved performance on the cognitive tests and vascular reactivity measure compared to following the control drink. It was thought this could be due to increased vaso-dilation and improving blood flow to the brain which was investigated in an extension to the project where a sample of individuals underwent brain imaging in an MRI scanner pre and post a blueberry and a control drink.

DETAILED DESCRIPTION:
The control drink was matched to the blueberry drink for other bioactive compounds which may have affected cognition, specifically sugars and vitamin C. Volunteers were healthy, not on any medication, without high blood pressure, high cholesterol, high BMI, diabetes or other medical conditions. Older adults were aged 61-75 years and younger adults 18-26 years.

Blood and urine samples will be analysed for flavonoid levels and Brain Derived Neurotrophic Factor, a biomarker of memory and learning, flavonoids may lead to increased BDNF production through the ERK-CREB-BDNF pathway.

Flavonoids may also increase nitric oxide production and improve the flexibility of the blood vessels hence the measure of vascular reactivity using the Digital Volume Pulse machine. This can lead to increased vaso-dilation and blood flow to the brain, therefore an fMRI study was carried out the investigate this using arterial spin labeling following acute blueberry supplementation compared to a control drink.

ELIGIBILITY:
Inclusion Criteria:

* No medical conditions
* Not taking any medication or supplements (or willing to stop taking supplements for duration of study)
* Not lactose intolerant
* Willing to give blood and urine samples
* Not partaking in frequent vigorous exercise
* Not suffering from or history of depression

Exclusion Criteria:

* On blood pressure medication, taking Aspirin or other blood thinning medication
* BMI > 30
* Cholesterol > 6
* Diabetes or other serious medical condition
* Lactose intolerant
* Any learning difficulty e.g. dyslexia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Cognitive function | pre drink, 2 hours and 5 hours post drink
  Extensive cognitive test battery including tasks measuring executive function such as updating, and memory tests such as free recall.

SECONDARY OUTCOMES:
Bioavailability and pharmacology | Pre drink and 1 hour post drink
  Flavonoid and BDNF levels in plasma and urine samples.
Vascular Reactivity | Pre and 1 hour post drink
  Measurements taken using Digital volume pulse equipment. Blood pressure also recorded.
Neuronal effects | Pre and 1 hours post drink
  Using fMRI to determine whether flavonoid supplementation leads to greater activation in brain regions associated with the cognitive abilities tested and to calculate cerebral blood flow before and after the blueberry compared to the control drink.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy PE Spencer, PhD, Principal Investigator — University of Reading; Laurie T Butler, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom